CLINICAL TRIAL: NCT05159609
Title: Closed Loop Auditory Stimulus in Sleep and epilepsY
Acronym: CLASSY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiff and Vale University Health Board (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 7796
Record Dates: First submitted 2021-11-25; First posted 2021-12-16 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Temporal Lobe Epilepsy
Keywords: Closed loop auditory stimulus; sleep; memory
MeSH Terms: conditions — Epilepsy, Temporal Lobe

STUDY DESIGN:
Intervention Model Description: Within subject comparison of stimulus and sham sessions
Who Masked: Participant
Masking Description: auditory stimulus was played at 0 or 50 decibels during sleep
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stim First (Active Comparator): Participants slept for one night while auditory sounds were played at specific points during slow wave sleep. At least one week later, an identical procedure occured with no acoustic sounds.
  Interventions: Device: Closed loop auditory stimulus
- Sham First (Sham Comparator): Participants slept for one night while no acoustic sounds were played. At least one week later, an identical procedure occured while acoustic sounds were played at specific points during slow wave sleep.
  Interventions: Device: Closed loop auditory stimulus

INTERVENTIONS:
Device: Closed loop auditory stimulus — 50ms of low volume pink noise delivered during slow wave sleep

SUMMARY:
This is a single-centre pilot study of a non-invasive auditory stimulation during sleep in participants with temporal lobe epilepsy.

DETAILED DESCRIPTION:
The primary objectives will be to pilot the use of home-based auditory stimulation during sleep in 10-20 participants with temporal lobe epilepsy using wireless devices.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is willing and able to give informed consent
2. Participant diagnosed with temporal lobe epilepsy
3. Will have had fewer than three generalized tonic clonic seizures per month in the last three months
4. Will be taking 3 or fewer anti-seizure medications.
5. Will have access to a computer or cellphone with an internet connection

Exclusion Criteria:

1. Abnormal hearing that cannot be corrected to normal overnight.
2. Abnormal vision that cannot be corrected to normal during the day.
3. Unwilling to abstain from caffeine, alcohol, daytime naps and extreme physical exercise in the 12 hours prior to the study.
4. Cannot read English
5. Engaged in night work in the previous 2 months
6. Any history of seizures triggered by music or sounds
7. Travelled across more than 2 time zones in the last 2 months
8. Prescribed/taking sleeping tablets other than clobazam
9. Cannabis use >4 joints/day.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Change in EEG waveform amplitude | 5 seconds after stimulus
  Does the acoustic sound delivery alter EEG waveform amplitude of slow wave sleep
Change in Serial Reaction Time Task memory test | Baseline and following day
  Does the delivery of acoustic sounds alter post-sleep preformance on the above task
Change in Paired Associates Learning memory test | Baseline and following day
  Does the delivery of acoustic sounds alter post-sleep preformance on the above task

CONTACTS AND LOCATIONS:
Overall Officials: Khalid Hamandi, MRCP/Phd, Principal Investigator — University Hospital of Wales/Cardiff University; Jennifer Roebber, PhD, Principal Investigator — University Hospital of Wales/Cardiff University
Locations (1):
- Cardiff and Vale UHW, Neurology department, ward C4, video-EEG monitoring unit, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymous sleeping-EEG and behavior scores can be shared with researchers.
Supporting Information: Analytic Code
Time Frame: Behavior tasks are available on Gitlab as a repository and can be shared on request